CLINICAL TRIAL: NCT00988117
Title: The Effects of the Rivastigmine Patch on Attention and Behavior in Parkinson's Disease With Dementia (PDD)
Brief Title: The Effects of the Rivastigmine Patch on Parkinson's Disease With Memory and/or Thinking Problems
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Bruce Miller, Director of the Memory & Aging Center, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA7 13D US45T
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Parkinsons Disease With Dementia; Parkinsons Disease With Mild to Moderate Memory and/or Thinking Problems
Keywords: PDD; Parkinson's Disease with Dementia; rivastigmine; rivastigmine patch; open label; Parkinson's Disease; Parkinsons Disease; memory; Exelon; Exelon Patch
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivastigmine Patch 9.5 cm2 (Experimental)
  Interventions: Drug: Rivastigmine Patch 9.5 cm2

INTERVENTIONS:
Drug: Rivastigmine Patch 9.5 cm2 — Subjects will be started on a 5cm2/24hr rivastigmine patch. After 4 weeks, the dose will be increased to a recommended target dose of 9.5cm2/24hr patch for 8 additional weeks.

SUMMARY:
This is an open-label study to investigate the effects of the rivastigmine patch on attention and behavior in Parkinson's disease when associated with memory and/or thinking problems. Rivastigmine (also sold under the name Exelon) is an FDA approved medication used for the treatment of mild to moderate Alzheimer's Disease (AD) and memory or thinking problems due to Parkinson's disease. Recently a rivastigmine patch was developed, which has shown similar effectiveness with fewer side effects and increased caregiver preference when compared to capsules. This is an open-label 12 week study where 15 subjects diagnosed with Parkinson's Disease who have mild to moderate memory and/or thinking complaints will be treated with the rivastigmine patch at UCSF. This study also analyzes the mechanism by which the rivastigmine patch works in people with Parkinson's disease and memory and/or thinking problems.

DETAILED DESCRIPTION:
Participation in this study requires four visits: a screening visit to ensure eligibility, an initial/baseline visit where the medication is distributed at a dosage lower than the optimal recommended dosage, a four week follow-up visit where the dosage of the medication is increased to the optimal amount, and a final twelve week follow up visit.

* In the screening visit the patient will undergo a neurological exam (including a review of their medical history and short physical exam), electrocardiogram ( a painless procedure that measures electrical activity of your heart), cognitive testing (such as memory and thinking tests), and a blood draw.
* At the Baseline/Initial visit the patient will receive a brief physical exam, additional cognitive testing, and an MRI scan. Afterwards, the study drug will be distributed.
* At the four week follow up visit the patient will be asked to do some abbreviated cognitive and neurological testing and the study drug will be re-distributed at the target dosage.
* At the final twelve week visit the patient will receive additional cognitive and neurological testing, and an MRI scan.
* Study compliance and adverse events will be reviewed every two weeks throughout the study, whether in person or over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Must meet research criteria for Parkinson's Disease with Dementia (PDD)
* Males and females, ages between 55 and 100
* Able to undergo psychometric testing
* Mini-Mental State Examination ≥ 21 and Clinical Dementia Rating < 2
* Reliable informant with frequent contact with patient

Exclusion Criteria:

* Non-English speaking, as cognitive tests will be in English
* Evidence of other neurological or psychiatric disorders which preclude diagnosis of PDD (including, but not limited to, stroke, any psychotic disorder, severe bipolar or unipolar depression, seizure disorder, or head injury with loss of consciousness) within the past year
* Concurrent treatment with any acetylcholinesterase inhibitors (including rivastigmine in pill or patch form), antipsychotic agents (excluding quetiapine in dosages of 150 mg and lower, abilify and geodon as these medications are commonly used in treatment of Parkinson's Disease (PD) psychosis and should not affect results of study), mood stabilizers (valproate or lithium) or benzodiazepines (other than temazepam or zolpidem)
* Positive urine drug screen or suspected alcohol or substance abuse within last 1 year
* Current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included
* Systolic blood pressure over 180 or less than 90 mm Hg. Diastolic blood pressure not greater than 105 or less than 50 mm Hg
* ECG is abnormal and judged to be clinically significant by the investigator
* Use of investigational drugs or participation in investigational drug studies within 30 days of screening
* Geriatric Depression Score score > 15/30
* Hachinski score > 4

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Miller, M.D., Principal Investigator — UCalifornia SF; Joel Kramer, PsyD, Study Director — UCalifornia SF
Locations (1):
- UCalifornia SF, San Francisco, California, United States

REFERENCES:
- [Result] Possin KL, Kang GA, Guo C, Fine EM, Trujillo AJ, Racine CA, Wilheim R, Johnson ET, Witt JL, Seeley WW, Miller BL, Kramer JH. Rivastigmine is associated with restoration of left frontal brain activity in Parkinson's disease. Mov Disord. 2013 Sep;28(10):1384-90. doi: 10.1002/mds.25575. Epub 2013 Jul 11. PMID 23847120
- See also: Information about the Memory & Aging Center at UCSF — http://memory.ucsf.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from UCSF movement disorders neurologists, regional Parkinson's Disease (PD) support group meetings and advertisements in PD newsletters between 4/2010 and 1/2011.
Groups:
- Rivastigmine: The Exelon patch (rivastigmine, Novartis International AG, Basel, Switzerland) was administered at a dosage of 4.6 mg/24 hours from baseline to week 4 and at 9.5 mg/24 hours from week 4 to 12.
Period: 4.6 mg/24 Hours From Baseline to Week 4
Arm/Group | Rivastigmine
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1
Period: 9.5 mg/24 Hours From Week 4 to 12
Arm/Group | Rivastigmine
Started | 14
Completed | 12
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours: The Exelon patch (rivastigmine, Novartis International AG, Basel, Switzerland) was administered at a dosage of 4.6 mg/24 hours from baseline to week 4 and at 9.5 mg/24 hours from week 4 to 12.
Arm/Group | Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Resting State Functional Activity Change From Baseline to 12 Weeks
Description: Fractional amplitude of low frequency fluctuations (fALFF) was used to measure brain activity. This metric is derived from task-free functional magnetic resonance imaging (fMRI) and represents the power of regional spontaneous and intrinsic brain activity at the local, voxel-wise level while the subject is at rest. More specifically, the amplitude of low-frequency fluctuations (ALFF) is the total power in the low-frequency range, and fALFF is calculated by dividing ALFF by the total power across all measurable frequencies. Whereas ALFF values increase near blood vessels and cerebrospinal fluid (CSF), likely due to pulsations in those areas, fALFF is less susceptible to artifactual signals. We measured change in these ratio scores post-treatment minus baseline and present in z-score units.
Time Frame: Baseline and 12 weeks
Population: All patients who completed the study were included.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours
Number analyzed (Participants) | 12
z-score
  left inferior frontal gyrus / premotor fALFF chang | 1.13 (1)
  left supplementary motor area fALFF change | .79 (1)
Statistical Analysis 1: Comparison: Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours; Each voxel's BOLD signal time series was detrended and transformed to the frequency domain. We divided the sum of the square roots across the 0.01-0.08 Hz range by that across the entire frequency range (0-0.25 Hz). fALFF group comparisons were evaluated using t-tests corrected for multiple comparisons. To determine if there were treatment-associated changes in brain activity, we compared voxel-wise fALFF in the patients at baseline to post-treatment; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — t-tests were statistically thresholded using the joint probability distribution method to correct for multiple comparisons, p < 0.01 for voxel height and p < 0.05 for cluster extent; A mask included only those regions where the patients showed abnormally low fALFF at either timepoint relative to a sample of 15 age-matched controls; Tscore = 5.19

2. Primary Outcome: Pre-post Change in Continuous Performance Test of Attention (Median Reaction Time)
Description: On the Continuous Performance Test (CPT), subjects press the spacebar quickly when they see a target image (a white star; 150 trials), and withhold response when they see a non-target image (5 randomly sampled white shapes; 150 trials). The inter-stimulus interval is randomly sampled from 1.5s, 2.5s, or 4s. Performance is measured by the median reaction time (milliseconds) on accurate target trials.
Time Frame: Baseline and 12 weeks
Population: Data were missing for two of the patients on the CPT post-treatment due to a computer error.
Measure: Median (Full Range); unit: milliseconds
Arm/Group | Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours
Number analyzed (Participants) | 10
milliseconds
  Baseline | 579 (108) [431 to 751]
  Post-treatment | 571 (108) [456 to 742]
Statistical Analysis 1: Comparison: Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours; correlation with left inferior frontal gyrus / premotor falff change; Test type: Superiority or Other; p < .01, Regression, Linear — This p-value was not adjusted for multiple comparisons; pearson's r correlation coefficient = -.82
Statistical Analysis 2: Comparison: Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours; correlation with left supplementary motor area falff change; Test type: Superiority or Other; p = .36, Regression, Linear — This p-value was not adjusted for multiple comparisons; pearson's correlation coefficient = -.35

3. Secondary Outcome: Pre-post Change in Montreal Cognitive Assessment
Description: The Montreal Cognitive Assessment (MoCA) was used as measure of global cognitive function. Total scores range from 0 (worst) to 30 (best).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours
Number analyzed (Participants) | 12
units on a scale
  Baseline | 23 (4.8)
  Post-treatment | 24.3 (4.7)
Statistical Analysis 1: Comparison: Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours; correlation with left premotor / inferior frontal gyri falff change; Test type: Superiority or Other; p = .58, Regression, Linear; pearson's r correlation = .18
Statistical Analysis 2: Comparison: Rivastigmine 4.6mg/24 Hours to 9.5mg/24 Hours; correlation with left supplementary motor area falff change; Test type: Superiority or Other; p = .41, Regression, Linear — This p-value was not adjusted for multiple comparisons; pearson's correlation coefficient = .26

ADVERSE EVENTS:
Groups:
- Rivastigmine 4.6mg/24 Hours: The Exelon patch (rivastigmine, Novartis International AG, Basel, Switzerland) was administered at a dosage of 4.6 mg/24 hours from baseline to week 4.
- Rivastigmine 9.5 mg/24 Hours: The Exelon patch was administered at a dosage of 9.5 mg/24 hours from week 4 to 12.
Arm/Group | Rivastigmine 4.6mg/24 Hours | Rivastigmine 9.5 mg/24 Hours
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/15 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivastigmine 4.6mg/24 Hours (N=15) | Rivastigmine 9.5 mg/24 Hours (N=14)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) — 1 subject dropped out of the study due to complaints of lightheadedness
gastrointestinal distress (Gastrointestinal disorders) | 0 (0) | 2 (2) — 2 subjects dropped out of the study due to reports of gastrointestinal distress

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No